CLINICAL TRIAL: NCT02249182
Title: A Phase 2, Open-Label, Multicenter, Multi-cohort Study to Investigate the Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed Dose Combination +/- Ribavirin in Adolescents and Children With Chronic HCV-Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed Dose Combination +/- Ribavirin in Adolescents and Children With Chronic HCV-Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1116; 2014-003578-17 (EudraCT Number)
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2019-03

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 12 to < 18 Years Old (Experimental): Participants between 12 to < 18 years of age weighing ≥ 45 kg will receive LDV/SOF FDC (90/400 mg tablet or 4 x 22.5 mg/100 mg tablets or 8 x 11.25/50 mg granules based on swallowability assessment during screening).
  Treatment duration will be dependent on HCV genotype, prior treatment experience, cirrhosis status, and country of enrollment.
  United Kingdom:
  * HCV genotypes (GT) 1, 4, 5, or 6 treatment-naive (TN) with or without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 treatment-experienced (TE) without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE with cirrhosis = LDV/SOF 24 weeks
  * HCV GT 3 TE with or without cirrhosis = LDV/SOF+RBV 24 weeks
  United States/Australia/New Zealand:
  * HCV GT 1, 4, 5, or 6 TN with or without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1 TE with cirrhosis = LDV/SOF 24 weeks
  * HCV GT 4, 5, or 6 TE with cirrhosis = LDV/SOF 12 weeks
  Interventions: Drug: LDV/SOF; Drug: RBV
- 6 to < 12 Years Old (Experimental): Participants between 6 to < 12 years of age weighing ≥ 17 kg and < 45 kg will receive LDV/SOF FDC (45/200 mg as 2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules based on swallowability assessment during screening).
  Treatment duration will be dependent on HCV genotype, prior treatment experience, cirrhosis status, and country of enrollment.
  United Kingdom:
  * HCV GT 1, 4, 5, or 6 TN with or without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE with cirrhosis = LDV/SOF 24 weeks
  * HCV GT 3 TE with or without cirrhosis = LDV/SOF+RBV 24 weeks
  United States/Australia/New Zealand:
  * HCV GT 1, 4, 5, or 6 TN with or without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1 TE with cirrhosis = LDV/SOF 24 weeks
  * HCV GT 4, 5, or 6 TE with cirrhosis = LDV/SOF 12 weeks
  Interventions: Drug: LDV/SOF; Drug: RBV
- 3 to < 6 Years Old (Experimental): Participants between 3 to < 6 years of age weighing ≥ 17 kg will receive LDV/SOF FDC (45/200 mg granules as 4 x 11.25/50 mg packets) and participants weighing < 17 kg will receive LDV/SOF FDC (33.75/150 mg oral granules as 3 x 11.25/50 mg packets).
  Treatment duration will be dependent on HCV genotype, prior treatment experience, cirrhosis status, and country of enrollment.
  United Kingdom:
  * HCV GT 1, 4, 5, or 6 TN with or without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE with cirrhosis = LDV/SOF 24 weeks
  * HCV GT 3 TE with or without cirrhosis = LDV/SOF+RBV 24 weeks
  United States/Australia/New Zealand:
  * HCV GT 1, 4, 5, or 6 TN with or without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1, 4, 5, or 6 TE without cirrhosis = LDV/SOF 12 weeks
  * HCV GT 1 TE with cirrhosis = LDV/SOF 24 weeks
  * HCV GT 4, 5, or 6 TE with cirrhosis = LDV/SOF 12 weeks
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF FDC administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — Ribavirin (RBV) oral solution or capsules will be administered orally in a divided daily dose based on weight
  Other Names: REBETOL®

SUMMARY:
The primary objective of the PK Lead-in Phase of the study is to evaluate the steady state pharmacokinetics (PK) and confirm the dose of ledipasvir/sofosbuvir (LDV/SOF) fixed dose combination (FDC) in hepatitis C virus (HCV)-infected pediatric participants. The PK Lead-in Phase will also evaluate the safety, tolerability, and antiviral activity of 10 days of dosing of LDV/SOF FDC in HCV-infected pediatric participants.

The Treatment Phase will be initiated by age cohort after confirmation of age-appropriate LDV/SOF FDC dosage levels. Participants from the PK Lead-in Phase will immediately rollover into the Treatment Phase with no interruption of study drug administration. The primary objective of the Treatment Phase is to evaluate the antiviral efficacy, safety, and tolerability of LDV/SOF FDC +/- ribavirin (RBV) for 12 or 24 weeks in pediatric participants with HCV.

During screening, participants will receive placebo to match LDV/SOF FDC to assess ability to swallow tablets.

ELIGIBILITY:
Key Inclusion Criteria:

* Consent of parent or legal guardian required
* Chronic HCV infection
* Screening laboratory values within defined thresholds

Key Exclusion Criteria:

* History of clinically significant illness or any other medical disorder that may interfere with individual's treatment, assessment or compliance with the protocol.
* Co-infection with HIV, acute hepatitis A virus, or hepatitis B virus
* Clinical hepatic decompensation (i.e., ascites, encephalopathy or variceal hemorrhage)
* Pregnant or nursing females
* Known hypersensitivity to study medication
* Use of any prohibited concomitant medications as within 28 days of the Day 1 visit

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 226 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (31):
- United States (23):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Morgantown, West Virginia
- Australia (3):
  - Newcastle, New South Wales
  - Westmead, New South Wales
  - Parkville, Victoria
- Auckland, New Zealand
- United Kingdom (4):
  - Birmingham, England
  - Leeds, England
  - London, England
  - Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Kirby B, German P, Kanwar B, Ni L, Lakatos I, Ling J, Mathias A. Pharmacokinetics of Once-Daily Sofosbuvir and Ledipasvir/Sofosbuvir in HCV-Infected Adolescents. Hepatology 2015;62 (S1): 1040A-1041A
- [Result] Garrison KL, Mathias A, Kersey K, Kanwar B, Ni L, Jain A, et al. Pharmacokinetics of Once-Daily Sofosbuvir and Ledipasvir/Sofosbuvir in HCV-Infected Pediatrics Aged 6 to < 12 Years Old. Hepatology 2016;64 (S1): 436A
- [Result] Schwarz K, Murray KF, Rosenthal P, Bansal S, Lin CH, Ni L, et al. High Rates of SVR12 in Adolescents Treated with the Combination of Ledipasvir/Sofosbuvir. J Hepatol 2016; 64 (2): S184-S185
- [Result] K.F. Murray, W. Balistreri, S. Bansal, S. Whitworth, H. Evans, R.P. Gonzalez-Peralta, et al. Ledipasvir/sofosbuvir ± ribavirin for 12 or 24 weeks is safe and effective in children 6-11 years old with chronic hepatitis C infection. J Hepatol 2017;66: S33-S62
- [Result] Balistreri WF, Murray KF, Rosenthal P, Bansal S, Lin CH, Kersey K, Massetto B, Zhu Y, Kanwar B, German P, Svarovskaia E, Brainard DM, Wen J, Gonzalez-Peralta RP, Jonas MM, Schwarz K. The safety and effectiveness of ledipasvir-sofosbuvir in adolescents 12-17 years old with hepatitis C virus genotype 1 infection. Hepatology. 2017 Aug;66(2):371-378. doi: 10.1002/hep.28995. Epub 2017 Jun 19. PMID 27997679
- [Result] Younossi ZM, Stepanova M, Balistreri W, Schwarz K, Murray KF, Rosenthal P, Bansal S, Hunt S. Health-related Quality of Life in Adolescent Patients With Hepatitis C Genotype 1 Treated With Sofosbuvir and Ledipasvir. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):112-116. doi: 10.1097/MPG.0000000000001754. PMID 28957984
- [Result] Begley R, Meng A, Massetto B, Shao J, Ling J, and Mathias A. Pharmacokinetics of Once Daily Sofosbuvir or Ledipasvir/Sofosbuvir in HCV-Infected Pediatrics Aged 3 to <6 Years Old. Hepatology 2018;68 (S1): 582A.
- [Result] Schwarz KB, Rosenthal P, Murray KF, Honegger JR, Hardikar W, Hague R, et al. Ledipasvir/Sofosbuvir for 12 Weeks Is Safe and Effective in Children 3 to <6 Years Old with Chronic Hepatitis C Virus Infection. Hepatology 2018;68 (S1): 116A-117A.
- [Result] Murray KF, Balistreri WF, Bansal S, Whitworth S, Evans HM, Gonzalez-Peralta RP, Wen J, Massetto B, Kersey K, Shao J, Garrison KL, Parhy B, Brainard DM, Arnon R, Gillis LA, Jonas MM, Lin CH, Narkewicz MR, Schwarz K, Rosenthal P. Safety and Efficacy of Ledipasvir-Sofosbuvir With or Without Ribavirin for Chronic Hepatitis C in Children Ages 6-11. Hepatology. 2018 Dec;68(6):2158-2166. doi: 10.1002/hep.30123. Epub 2018 Nov 17. PMID 30070726
- [Derived] Schwarz KB, Rosenthal P, Murray KF, Honegger JR, Hardikar W, Hague R, Mittal N, Massetto B, Brainard DM, Hsueh CH, Shao J, Parhy B, Narkewicz MR, Rao GS, Whitworth S, Bansal S, Balistreri WF. Ledipasvir-Sofosbuvir for 12 Weeks in Children 3 to <6 Years Old With Chronic Hepatitis C. Hepatology. 2020 Feb;71(2):422-430. doi: 10.1002/hep.30830. Epub 2019 Aug 19. PMID 31220349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, United Kingdom, Australia, and New Zealand. The first participant was screened on 05 November 2014. The last study visit occurred on 24 August 2018.
Pre-assignment Details: 240 participants were screened.
Groups:
- 12 to < 18 Years Old - LDV/SOF 12 Weeks: Participants 12 to < 18 years of age with hepatitis C virus (HCV) genotype 1 treatment-naive (TN) with or without cirrhosis or treatment-experienced (TE) without cirrhosis received ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) 90/400 mg (1 x 90/400 mg tablet or 4 x 22.5/100 mg tablets) once daily for 12 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
- 6 to < 12 Years Old - LDV/SOF 12 Weeks: Participants 6 to < 12 years of age with HCV genotypes 1 or 4 TN with or without cirrhosis or HCV genotype 1 TE without cirrhosis received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily for 12 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
- 6 to < 12 Years Old - LDV/SOF 24 Weeks: Participants 6 to < 12 years of age with HCV genotype 1 TE with cirrhosis received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily for 24 weeks.
- 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks: Participants 6 to < 12 years of age with HCV genotype 3 TE without cirrhosis received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily + ribavirin (RBV) capsules or oral solution (dose depending on weight) for 24 weeks.
- 3 to < 6 Years Old - LDV/SOF 12 Weeks: Participants 3 to < 6 years of age with HCV genotypes 1 or 4 TN without cirrhosis received LDV/SOF FDC (weight ≥ 17 kg: 45/200 mg granules; weight < 17 kg: 33.75/150 mg granules) once daily for 12 weeks. Participants participating in the PK Lead-in Phase immediately rolled over into the Treatment Phase without interruption to study drug administration.
Period: PK Lead-In Phase
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Started | 10 | 12 | 0 | 0 | 17
Completed | 10 | 12 | 0 | 0 | 17
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Started | 100 (90 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 89 (77 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 1 (1 participant enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 2 (2 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.) | 34 (17 participants enrolled directly into the Treatment Phase, without entering the PK Lead-In Phase.)
Completed | 96 | 89 | 1 | 2 | 34
Not Completed | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
Groups:
- 12 to < 18 Years Old - LDV/SOF 12 Weeks: Participants 12 to < 18 years of age with HCV genotype 1 TN with or without cirrhosis or HCV genotype 1 TE without cirrhosis received LDV/SOF FDC 90/400 mg (1 x 90/400 mg tablet or 4 x 22.5/100 mg tablets) once daily for 12 weeks.
- 6 to < 12 Years Old - LDV/SOF 12 Weeks: Participants 6 to < 12 years of age with HCV genotypes 1 or 4 TN with or without cirrhosis or HCV genotype 1 TE without cirrhosis received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily for 12 weeks.
- 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks: Participants 6 to < 12 years of age with HCV genotype 3 TE without cirrhosis received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily + ribavirin capsules or oral solution (dose depending on weight) for 24 weeks.
- 3 to < 6 Years Old - LDV/SOF 12 Weeks: Participants 3 to < 6 years of age with HCV genotypes 1 or 4 TN without cirrhosis received LDV/SOF FDC (weight ≥ 17 kg: 45/200 mg granules; weight < 17 kg: 33.75/150 mg granules) once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks | Total
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.7) | 9 (1.6) | 11 (NA) — Standard deviation of a single sample is undefined. | 9 (2.8) | 4 (0.7) | 11 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 36 | 1 | 1 | 24 | 125
  Male | 37 | 53 | 0 | 1 | 10 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 91 | 70 | 1 | 2 | 27 | 191
  Black or African American | 7 | 7 | 0 | 0 | 1 | 15
  Other | 0 | 5 | 0 | 0 | 4 | 9
  Asian | 2 | 5 | 0 | 0 | 2 | 9
  Native Hawaiian or Pacific Islander | 0 | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 0 | 0 | 6 | 28
  Not Hispanic or Latino | 85 | 75 | 1 | 2 | 28 | 191
  Not Disclosed | 2 | 5 | 0 | 0 | 0 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 0 | 4 | 0 | 0 | 0 | 4
  United States | 91 | 70 | 0 | 0 | 29 | 190
  United Kingdom | 1 | 9 | 0 | 2 | 3 | 15
  Australia | 8 | 6 | 1 | 0 | 2 | 17
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 100 | 87 | 1 | 0 | 33 | 221
  Genotype 3 | 0 | 0 | 0 | 2 | 0 | 2
  Genotype 4 | 0 | 2 | 0 | 0 | 1 | 3
Cirrhosis Status [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 1 | 0 | 0 | 3
  No | 43 | 33 | 0 | 2 | 14 | 92
  Unknown | 56 | 55 | 0 | 0 | 20 | 131
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 24 | 23 | 0 | 0 | 10 | 57
    CT | 53 | 53 | 0 | 2 | 16 | 124
    TT | 23 | 12 | 1 | 0 | 6 | 42
    Missing | 0 | 1 | 0 | 0 | 2 | 3
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 45 | 37 | 0 | 1 | 15 | 98
  ≥ 800,000 IU/mL | 55 | 52 | 1 | 1 | 19 | 128
Prior Treatment Experience [Count of Participants; unit: Participants]
  Treatment-Naive | 80 | 72 | 0 | 0 | 34 | 186
  Treatment-Experienced | 20 | 17 | 1 | 2 | 0 | 40

OUTCOME MEASURES:

1. Primary Outcome: For Participants in the PK Lead-in Phase, Pharmacokinetic (PK) Parameter: AUCtau of GS-331007 (Metabolite of SOF), LDV, and SOF
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Cohorts 1 and 2 (6 to < 18 years of age): predose, 0.5, 1, 2, 3, 4, 5, 8, and 12 hours postdose on Day 10; Cohort 3 (3 to < 6 years of age): predose, 0.5, 2, 4, 8, and 12 hours postdose on Day 10
Population: Intensive PK Analysis Set included all participants in the PK lead-in phase who received at least 1 dose of study drug and for whom at least 1 nonmissing PK concentration value, during the intensive sampling period, was reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- PK Lead-in: 12 to < 18 Years Old - LDV/SOF 12 Weeks: Participants 12 to < 18 years of age weighing ≥ 45 kg received LDV/SOF FDC 90/400 mg (1 x 90/400 mg tablet or 4 x 22.5/100 mg tablets) once daily for 12 weeks.
- PK Lead-in: 6 to < 12 Years Old - LDV/SOF 12 Weeks: Participants 6 to < 12 years of age weighing ≥ 17 kg and < 45 kg received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily for 12 weeks.
- PK Lead-in: 3 to < 6 Years Old - LDV/SOF 12 Weeks: Participants 3 to < 6 years of age received LDV/SOF FDC (weight ≥ 17 kg: 45/200 mg granules; weight < 17 kg: 33.75/150 mg granules) once daily for 12 weeks.
Arm/Group | PK Lead-in: 12 to < 18 Years Old - LDV/SOF 12 Weeks | PK Lead-in: 6 to < 12 Years Old - LDV/SOF 12 Weeks | PK Lead-in: 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 10 | 10 | 13
h*ng/mL
  GS-331007 (metabolite of SOF) | 12682.5 (1732.66) | 8210.3 (2542.42) | 11688.9 (3400.79)
  LDV | 10202.4 (5196.49) | 7288.3 (4547.33) | 9316.3 (3280.51)
  SOF: number analyzed (Participants) | 10 | 9 | 3
  SOF | 2175.7 (578.92) | 1754.4 (419.18) | 2495.2 (412.64)
Statistical Analysis 1: Comparison: PK Lead-in: 12 to < 18 Years Old - LDV/SOF 12 Weeks; AUCtau of GS-331007 for the 12 to < 18 Years old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — Equivalence was determined if the 90% confidence intervals (CI) were within the predefined equivalence boundaries of 50% to 200% for all age groups; Percentage Geometric Mean Ratio = 105.20, 90% CI 2-sided [90.61 to 122.13]
Statistical Analysis 2: Comparison: PK Lead-in: 6 to < 12 Years Old - LDV/SOF 12 Weeks; AUCtau of GS-331007 for the 6 to < 12 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — Equivalence was determined if the 90% CIs were within the predefined equivalence boundaries of 50% to 200% for all age groups; Percentage Geometric Mean Ratio = 65.76, 90% CI 2-sided [56.62 to 76.37]
Statistical Analysis 3: Comparison: PK Lead-in: 3 to < 6 Years Old - LDV/SOF 12 Weeks; AUCtau of GS-331007 for the 3 to < 6 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 94.08, 90% CI 2-sided [82.51 to 107.27]
Statistical Analysis 4: Comparison: PK Lead-in: 12 to < 18 Years Old - LDV/SOF 12 Weeks; AUCtau of LDV for the 12 to < 18 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 127.18, 90% CI 2-sided [94.89 to 170.45]
Statistical Analysis 5: Comparison: PK Lead-in: 6 to < 12 Years Old - LDV/SOF 12 Weeks; AUCtau of LDV for the 6 to < 12 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 82.25, 90% CI 2-sided [61.34 to 110.30]
Statistical Analysis 6: Comparison: PK Lead-in: 3 to < 6 Years Old - LDV/SOF 12 Weeks; AUCtau of LDV for the 3 to < 6 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 120.46, 90% CI 2-sided [93.18 to 155.73]
Statistical Analysis 7: Comparison: PK Lead-in: 12 to < 18 Years Old - LDV/SOF 12 Weeks; AUCtau of SOF for the 12 to < 18 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 159.88, 90% CI 2-sided [137.89 to 185.37]
Statistical Analysis 8: Comparison: PK Lead-in: 6 to < 12 Years Old - LDV/SOF 12 Weeks; AUCtau of SOF for the 6 to < 12 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 129.48, 90% CI 2-sided [110.79 to 151.32]
Statistical Analysis 9: Comparison: PK Lead-in: 3 to < 6 Years Old - LDV/SOF 12 Weeks; AUCtau of SOF for the 3 to < 6 Years Old group in the PK Lead-in Phase was compared against historical data collected in adult Phase 2/3 studies; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Percentage Geometric Mean Ratio = 187.76, 90% CI 2-sided [143.41 to 245.82]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event During the PK Lead-in Phase or the Treatment Phase
Time Frame: Up to 24 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- 12 to < 18 Years Old - LDV/SOF 12 Weeks: Participants 12 to < 18 years of age with HCV genotype 1 TN with or without cirrhosis or TE without cirrhosis received LDV/SOF FDC 90/400 mg (1 x 90/400 mg tablet or 4 x 22.5/100 mg tablets) once daily for 12 weeks.
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
percentage of participants | 0 | 0 | 0 | 0 | 2.9

3. Secondary Outcome: For Participants in the PK Lead-in Phase, Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12
Population: Participants who were enrolled in the PK lead-in phase with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PK Lead-in: 12 to < 18 Years Old - LDV/SOF 12 Weeks | PK Lead-in: 6 to < 12 Years Old - LDV/SOF 12 Weeks | PK Lead-in: 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 10 | 12 | 17
log10 IU/mL
  Change at Week 1 | -4.34 (0.621) | -4.29 (0.518) | -4.32 (0.616)
  Change at Week 2: number analyzed (Participants) | 10 | 12 | 15
  Change at Week 2 | -4.71 (0.651) | -4.55 (0.636) | -4.87 (0.724)
  Change at Week 4: number analyzed (Participants) | 10 | 12 | 16
  Change at Week 4 | -4.73 (0.667) | -4.75 (0.702) | -4.92 (0.715)
  Change at Week 8: number analyzed (Participants) | 10 | 12 | 16
  Change at Week 8 | -4.73 (0.667) | -4.76 (0.710) | -4.92 (0.715)
  Change at Week 12: number analyzed (Participants) | 10 | 12 | 16
  Change at Week 12 | -4.73 (0.667) | -4.76 (0.710) | -4.92 (0.715)

4. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event During the PK Lead-in Phase
Time Frame: Up to Day 10
Population: Participants who were enrolled in the PK lead-in phase were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | PK Lead-in: 12 to < 18 Years Old - LDV/SOF 12 Weeks | PK Lead-in: 6 to < 12 Years Old - LDV/SOF 12 Weeks | PK Lead-in: 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 10 | 12 | 17
percentage of participants | 0 | 0 | 5.9

5. Secondary Outcome: For the Treatment Phase, Percentage of Participants With Sustained Virologic Response (SVR) at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
percentage of participants | 98.0 [93.0 to 99.8] | 98.9 [93.9 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 97.1 [84.7 to 99.9]

6. Secondary Outcome: For the Treatment Phase, Percentage of Participants With SVR at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < LLOQ at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
percentage of participants | 98.0 [93.0 to 99.8] | 98.9 [93.9 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 97.1 [84.7 to 99.9]

7. Secondary Outcome: For the Treatment Phase, Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
percentage of participants | 98.0 [93.0 to 99.8] | 98.9 [93.9 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 97.1 [84.7 to 99.9]

8. Secondary Outcome: For the Treatment Phase, Percentage of Participants Experiencing Viral Breakthrough
Description: Viral breakthrough was defined as having confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment.
Time Frame: Up to 24 weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
percentage of participants | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: For the Treatment Phase, Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as having confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
percentage of participants | 0 | 1.1 | 0 | 0 | 0

10. Secondary Outcome: For the Treatment Phase, Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only)
Population: Participants in the Full Analysis Set with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Change at Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 98 | 85 | 1 | 2 | 34
  Change at Week 1 | -4.34 (0.634) | -4.27 (0.592) | -4.30 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) | -4.25 (0.505)
  Change at Week 2: number analyzed (Participants) | 99 | 88 | 1 | 2 | 32
  Change at Week 2 | -4.74 (0.585) | -4.73 (0.544) | -5.09 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) | -4.80 (0.628)
  Change at Week 4: number analyzed (Participants) | 100 | 89 | 1 | 2 | 33
  Change at Week 4 | -4.84 (0.557) | -4.87 (0.592) | -5.09 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) | -4.85 (0.628)
  Change at Week 8: number analyzed (Participants) | 99 | 89 | 1 | 2 | 33
  Change at Week 8 | -4.85 (0.556) | -4.89 (0.597) | -5.09 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) | -4.86 (0.633)
  Change at Week 12: number analyzed (Participants) | 99 | 89 | 1 | 2 | 33
  Change at Week 12 | -4.85 (0.556) | -4.89 (0.597) | -5.09 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) | -4.86 (0.633)
  Change at Week 16: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 16 |  |  | -5.09 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) |
  Change at Week 20: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 20 |  |  | -5.09 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) |
  Change at Week 24: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 24 |  |  | -5.09 (NA) — Standard deviation of a single sample is undefined. | -4.54 (0.308) |

11. Secondary Outcome: For the Treatment Phase, Percentage of Participants With HCV RNA < LLOQ While On Treatment
Time Frame: Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only)
Population: Participants in the Full Analysis Set with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
percentage of participants
  Week 1 | 40.0 [30.3 to 50.3] | 30.3 [21.0 to 41.0] | 0 [0.0 to 97.5] | 100.0 [15.8 to 100.0] | 29.4 [15.1 to 47.5]
  Week 2: number analyzed (Participants) | 100 | 89 | 1 | 2 | 33
  Week 2 | 75.0 [65.3 to 83.1] | 71.9 [61.4 to 80.9] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 78.8 [61.1 to 91.0]
  Week 4: number analyzed (Participants) | 100 | 89 | 1 | 2 | 33
  Week 4 | 97.0 [91.5 to 99.4] | 96.6 [90.5 to 99.3] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 97.0 [84.2 to 99.9]
  Week 8: number analyzed (Participants) | 99 | 89 | 1 | 2 | 33
  Week 8 | 100.0 [96.3 to 100.0] | 100.0 [95.9 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [89.4 to 100.0]
  Week 12: number analyzed (Participants) | 99 | 89 | 1 | 2 | 33
  Week 12 | 100.0 [96.3 to 100.0] | 100.0 [95.9 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [89.4 to 100.0]
  Week 16: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Week 16 |  |  | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] |
  Week 20: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Week 20 |  |  | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] |
  Week 24: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Week 24 |  |  | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] |

12. Secondary Outcome: For the Treatment Phase, Percentage of Participants With Alanine Aminotransferase (ALT) Normalization
Description: ALT normalization was defined as ALT > the upper limit of normal (ULN) at baseline and ALT ≤ ULN at each visit.
Time Frame: Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only), and Posttreatment Week 4
Population: Participants in the Full Analysis Set with ALT > ULN at Baseline with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 49 | 72 | 1 | 2 | 27
percentage of participants
  Week 1: number analyzed (Participants) | 47 | 70 | 1 | 2 | 27
  Week 1 | 72.3 | 75.7 | 0 | 50.0 | 63.0
  Week 2: number analyzed (Participants) | 49 | 66 | 1 | 2 | 25
  Week 2 | 89.8 | 84.8 | 0 | 50.0 | 84.0
  Week 4: number analyzed (Participants) | 48 | 72 | 1 | 2 | 25
  Week 4 | 93.8 | 93.1 | 0 | 100.0 | 96.0
  Week 8: number analyzed (Participants) | 46 | 71 | 1 | 2 | 25
  Week 8 | 91.3 | 90.1 | 0 | 100.0 | 92.0
  Week 12: number analyzed (Participants) | 45 | 67 | 1 | 2 | 24
  Week 12 | 93.3 | 95.5 | 100.0 | 100.0 | 91.7
  Week 16: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Week 16 |  |  | 100.0 | 100.0 |
  Week 20: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Week 20 |  |  | 100.0 | 100.0 |
  Week 24: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Week 24 |  |  | 100.0 | 100.0 |
  Posttreatment Week 4: number analyzed (Participants) | 41 | 62 | 0 | 2 | 23
  Posttreatment Week 4 | 90.2 | 98.4 |  | 100.0 | 91.3

13. Secondary Outcome: For the Treatment Phase, Change From Baseline in Height
Time Frame: Baseline; Weeks 1, 2, 4, 8, 12, 16 (24 Week groups only), 20 (24 Week groups only), and 24 (24 Week groups only), and Posttreatment Weeks 4, 12, and 24
Population: Participants in the Safety Analysis Set with available data were analyzed. Participants from the 12 Weeks groups were not analyzed for Change at Weeks 16, 20, and 24 because they were only treated for 12 weeks.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
centimeters
  Change at Week 1: number analyzed (Participants) | 97 | 85 | 1 | 2 | 34
  Change at Week 1 | 0.1 (0.68) | 0.1 (0.83) | 0.3 (NA) — Standard deviation of a single sample is undefined. | 0.7 (1.13) | 0.2 (1.24)
  Change at Week 2: number analyzed (Participants) | 97 | 86 | 1 | 2 | 32
  Change at Week 2 | 0.0 (0.70) | 0.3 (0.73) | 0.5 (NA) — Standard deviation of a single sample is undefined. | 0.5 (0.85) | 0.3 (0.72)
  Change at Week 4: number analyzed (Participants) | 98 | 87 | 1 | 2 | 33
  Change at Week 4 | 0.1 (0.84) | 0.5 (0.79) | 1.2 (NA) — Standard deviation of a single sample is undefined. | 0.6 (0.92) | 0.7 (0.79)
  Change at Week 8: number analyzed (Participants) | 98 | 88 | 1 | 2 | 33
  Change at Week 8 | 0.4 (1.04) | 0.8 (0.79) | 1.3 (NA) — Standard deviation of a single sample is undefined. | 0.8 (0.92) | 1.0 (0.82)
  Change at Week 12: number analyzed (Participants) | 92 | 84 | 1 | 2 | 31
  Change at Week 12 | 0.5 (1.10) | 1.3 (0.83) | 2.1 (NA) — Standard deviation of a single sample is undefined. | 1.1 (1.41) | 1.6 (0.98)
  Change at Week 16: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 16 |  |  | 3.2 (NA) — Standard deviation of a single sample is undefined. | 1.4 (1.06) |
  Change at Week 20: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 20 |  |  | 4.3 (NA) — Standard deviation of a single sample is undefined. | 1.6 (0.85) |
  Change at Week 24: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 24 |  |  | 4.3 (NA) — Standard deviation of a single sample is undefined. | 2.5 (1.48) |
  Change at Posttreatment Week 4: number analyzed (Participants) | 97 | 89 | 1 | 2 | 34
  Change at Posttreatment Week 4 | 0.8 (1.46) | 1.8 (1.04) | 4.3 (NA) — Standard deviation of a single sample is undefined. | 2.4 (1.27) | 2.1 (1.13)
  Change at Posttreatment Week 12: number analyzed (Participants) | 96 | 87 | 1 | 2 | 34
  Change at Posttreatment Week 12 | 1.2 (1.82) | 2.7 (0.97) | 5.0 (NA) — Standard deviation of a single sample is undefined. | 3.4 (1.56) | 3.3 (1.18)
  Change at Posttreatment Week 24: number analyzed (Participants) | 95 | 88 | 1 | 2 | 34
  Change at Posttreatment Week 24 | 1.8 (2.31) | 4.1 (1.39) | 7.6 (NA) — Standard deviation of a single sample is undefined. | 5.6 (0.85) | 4.7 (1.31)

14. Secondary Outcome: For the Treatment Phase, Change From Baseline in Weight
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 100 | 89 | 1 | 2 | 34
kilograms
  Change at Week 1: number analyzed (Participants) | 98 | 86 | 1 | 2 | 34
  Change at Week 1 | 0.1 (1.00) | 0.3 (0.51) | -0.5 (NA) — Standard deviation of a single sample is undefined. | 0.3 (1.34) | 0.1 (0.39)
  Change at Week 2: number analyzed (Participants) | 97 | 87 | 1 | 2 | 33
  Change at Week 2 | 0.3 (1.11) | 0.4 (0.54) | 0.0 (NA) — Standard deviation of a single sample is undefined. | 0.3 (1.77) | 0.2 (0.44)
  Change at Week 4: number analyzed (Participants) | 98 | 89 | 1 | 2 | 33
  Change at Week 4 | 0.4 (1.44) | 0.5 (0.64) | 0.5 (NA) — Standard deviation of a single sample is undefined. | 0.7 (1.91) | 0.3 (0.64)
  Change at Week 8: number analyzed (Participants) | 98 | 89 | 1 | 2 | 33
  Change at Week 8 | 0.5 (1.90) | 0.8 (0.84) | 1.3 (NA) — Standard deviation of a single sample is undefined. | 0.6 (2.33) | 0.5 (0.66)
  Change at Week 12: number analyzed (Participants) | 92 | 84 | 1 | 2 | 31
  Change at Week 12 | 0.6 (2.32) | 1.1 (1.27) | 2.1 (NA) — Standard deviation of a single sample is undefined. | 0.9 (2.90) | 0.6 (0.70)
  Change at Week 16: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 16 |  |  | 1.6 (NA) — Standard deviation of a single sample is undefined. | 1.2 (3.68) |
  Change at Week 20: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 20 |  |  | 2.2 (NA) — Standard deviation of a single sample is undefined. | 1.8 (3.96) |
  Change at Week 24: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0
  Change at Week 24 |  |  | 3.1 (NA) — Standard deviation of a single sample is undefined. | 2.4 (3.68) |
  Change at Posttreatment Week 4: number analyzed (Participants) | 97 | 89 | 1 | 2 | 34
  Change at Posttreatment Week 4 | 0.9 (2.70) | 1.4 (1.48) | 1.8 (NA) — Standard deviation of a single sample is undefined. | 2.2 (3.68) | 1.1 (1.09)
  Change at Posttreatment Week 12: number analyzed (Participants) | 96 | 89 | 1 | 2 | 34
  Change at Posttreatment Week 12 | 1.6 (3.48) | 2.1 (1.87) | 3.1 (NA) — Standard deviation of a single sample is undefined. | 3.7 (2.90) | 1.2 (0.93)
  Change at Posttreatment Week 24: number analyzed (Participants) | 95 | 89 | 1 | 2 | 34
  Change at Posttreatment Week 24 | 3.2 (4.38) | 3.5 (2.75) | 4.5 (NA) — Standard deviation of a single sample is undefined. | 5.7 (1.41) | 2.0 (1.57)

15. Secondary Outcome: For the Treatment Phase, Number of Male Participants With a Change From Baseline in Tanner Stage for Pubic Hair
Description: Tanner Stages is a scale that defines physical measurements of development based on external primary and secondary sex characteristics. It was used in this study to assess pubertal development with values ranging from Stage 1 (pre-pubertal characteristics) to Stage 5 (adult or mature characteristics). Any shifts (increase or decrease) in Tanner Stage from Baseline were analyzed and presented.
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Male participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- 12 to < 18 Years Old - LDV/SOF 12 Weeks: Male participants 12 to < 18 years of age received LDV/SOF FDC 90/400 mg (1 x 90/400 mg tablet or 4 x 22.5/100 mg tablets) once daily for 12 weeks.
- 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks: Male participants 6 to < 12 years of age received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily ± RBV capsules or oral solution (dose depending on weight) for 12 or 24 weeks.
- 3 to < 6 Years Old - LDV/SOF 12 Weeks: Male participants 3 to < 6 years of age received LDV/SOF FDC (weight ≥ 17 kg: 45/200 mg granules; weight < 17 kg: 33.75/150 mg granules) once daily for 12 weeks.
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 37 | 54 | 10
Participants
  End of Treatment: number analyzed (Participants) | 36 | 54 | 10
  End of Treatment: No Change | 35 | 52 | 10
  End of Treatment: Increase | 1 | 1 | 0
  End of Treatment: Decrease | 0 | 1 | 0
  Posttreatment Week 12: number analyzed (Participants) | 35 | 54 | 9
  Posttreatment Week 12: No Change | 32 | 51 | 9
  Posttreatment Week 12: Increase | 3 | 2 | 0
  Posttreatment Week 12: Decrease | 0 | 1 | 0
  Posttreatment Week 24: number analyzed (Participants) | 35 | 53 | 10
  Posttreatment Week 24: No Change | 28 | 48 | 9
  Posttreatment Week 24: Increase | 7 | 4 | 1
  Posttreatment Week 24: Decrease | 0 | 1 | 0

16. Secondary Outcome: For the Treatment Phase, Number of Male Participants With a Change From Baseline in Tanner Stage for Genitalia Development
Description: as for outcome 15
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Male participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 37 | 54 | 10
Participants
  End of Treatment: number analyzed (Participants) | 35 | 54 | 10
  End of Treatment: No Change | 34 | 52 | 10
  End of Treatment: Increase | 1 | 1 | 0
  End of Treatment: Decrease | 0 | 1 | 0
  Posttreatment Week 12: number analyzed (Participants) | 35 | 54 | 9
  Posttreatment Week 12: No Change | 33 | 50 | 9
  Posttreatment Week 12: Increase | 2 | 4 | 0
  Posttreatment Week 12: Decrease | 0 | 0 | 0
  Posttreatment Week 24: number analyzed (Participants) | 35 | 53 | 10
  Posttreatment Week 24: No Change | 29 | 47 | 10
  Posttreatment Week 24: Increase | 6 | 6 | 0
  Posttreatment Week 24: Decrease | 0 | 0 | 0

17. Secondary Outcome: For the Treatment Phase, Number of Female Participants With a Change From Baseline in Tanner Stage for Pubic Hair
Description: as for outcome 15
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Female participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- 12 to < 18 Years Old - LDV/SOF 12 Weeks: Female participants 12 to < 18 years of age received LDV/SOF FDC 90/400 mg (1 x 90/400 mg tablet or 4 x 22.5/100 mg tablets) once daily for 12 weeks.
- 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks: Female participants 6 to < 12 years of age received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily ± RBV capsules or oral solution (dose depending on weight) for 12 or 24 weeks.
- 3 to < 6 Years Old - LDV/SOF 12 Weeks: Female participants 3 to < 6 years of age received LDV/SOF FDC (weight ≥ 17 kg: 45/200 mg granules; weight < 17 kg: 33.75/150 mg granules) once daily for 12 weeks.
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 63 | 38 | 24
Participants
  End of Treatment: number analyzed (Participants) | 62 | 36 | 21
  End of Treatment: No Change | 52 | 34 | 21
  End of Treatment: Increase | 9 | 2 | 0
  End of Treatment: Decrease | 1 | 0 | 0
  Posttreatment Week 12: number analyzed (Participants) | 60 | 34 | 22
  Posttreatment Week 12: No Change | 45 | 31 | 22
  Posttreatment Week 12: Increase | 15 | 3 | 0
  Posttreatment Week 12: Decrease | 0 | 0 | 0
  Posttreatment Week 24: number analyzed (Participants) | 61 | 35 | 22
  Posttreatment Week 24: No Change | 40 | 27 | 22
  Posttreatment Week 24: Increase | 21 | 8 | 0
  Posttreatment Week 24: Decrease | 0 | 0 | 0

18. Secondary Outcome: For the Treatment Phase, Number of Female Participants With a Change From Baseline in Tanner Stage for Breast Development
Description: as for outcome 15
Time Frame: Baseline; End of Treatment (either Week 12 or 24), Posttreatment Week 12, and Posttreatment Week 24
Population: Female participants in the Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 63 | 38 | 24
Participants
  End of Treatment: number analyzed (Participants) | 62 | 36 | 21
  End of Treatment: No Change | 53 | 31 | 21
  End of Treatment: Increase | 8 | 5 | 0
  End of Treatment: Decrease | 1 | 0 | 0
  Posttreatment Week 12: number analyzed (Participants) | 60 | 34 | 22
  Posttreatment Week 12: No Change | 49 | 25 | 21
  Posttreatment Week 12: Increase | 11 | 8 | 1
  Posttreatment Week 12: Decrease | 0 | 1 | 0
  Posttreatment Week 24: number analyzed (Participants) | 61 | 35 | 22
  Posttreatment Week 24: No Change | 43 | 21 | 21
  Posttreatment Week 24: Increase | 18 | 14 | 1
  Posttreatment Week 24: Decrease | 0 | 0 | 0

19. Secondary Outcome: Acceptability of LDV/SOF Tablets as Measured by the Percentage of Participants Able/Unable to Swallow Placebo Tablet at Day 1
Description: Participants who were able/unable to swallow placebo tablets were assessed. Participants 12 to < 18 years old were first asked to perform the swallowability assessment using the 90/400 mg placebo tablet. If they were unable to swallow this, they were then asked to perform the swallowability assessment with 22.5/100 mg placebo tablets. Participants 6 to < 12 years old were to be assessed with the 22.5/100 mg placebo tablets. However, 8 participants were mistakenly assessed using the 90/400 mg placebo tablet.
Time Frame: Day 1
Population: Participants between 6 to <18 years old in the Safety Analysis Set who performed the swallowability assessment were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- 12 to < 18 Years Old - LDV/SOF 12 Weeks: Participants 12 to < 18 years of age received placebo to match LDV/SOF FDC to assess ability to swallow tablets on Day 1. They then received LDV/SOF FDC 90/400 mg (1 x 90/400 mg tablet or 4 x 22.5/100 mg tablets) once daily for 12 weeks.
- 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks: Participants 6 to < 12 years of age received placebo to match LDV/SOF FDC to assess ability to swallow tablets on Day 1. They then received LDV/SOF FDC 45/200 mg (2 x 22.5/100 mg tablets or 4 x 11.25/50 mg granules) once daily ± RBV capsules or oral solution (dose depending on weight) for 12 or 24 weeks.
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF±RBV 12 or 24 Weeks
Number analyzed (Participants) | 100 | 92
percentage of participants
  Able to Swallow 90/400 mg Placebo Tablet: number analyzed (Participants) | 100 | 8
  Able to Swallow 90/400 mg Placebo Tablet | 89.0 | 100.0
  Unable to Swallow 90/400 mg Placebo Tablet: number analyzed (Participants) | 100 | 8
  Unable to Swallow 90/400 mg Placebo Tablet | 11.0 | 0
  Able to Swallow 22.5/100 mg Placebo Tablet: number analyzed (Participants) | 11 | 84
  Able to Swallow 22.5/100 mg Placebo Tablet | 72.7 | 98.8
  Unable to Swallow 22.5/100 mg Placebo Tablet: number analyzed (Participants) | 11 | 84
  Unable to Swallow 22.5/100 mg Placebo Tablet | 27.3 | 1.2

20. Secondary Outcome: Acceptability of LDV/SOF Granules as Measured by Palatability at Day 1
Description: Participants who were dosed with granules were asked if they tasted the study drug. If they tasted it, then they were asked to provide a number from 0 to 100 to rate the taste of the study drug, with higher scores indicating better taste. Data was then summarized as percentage of participants choosing the following palatability categories: 1) Did not taste the study drug, 2) Tasted drug with score > 60 to 100, 3) Tasted drug with score 40 to 60, and 4) Tasted drug with score of 0 to < 40.
Time Frame: Day 1
Population: Participants between 3 to <6 years old in the Safety Analysis Set who performed the palatability test were analyzed.
Measure: Number; unit: percentage of participants
Groups:
- 3 to < 6 Years Old - LDV/SOF 12 Weeks: Participants 3 to < 6 years of age received LDV/SOF FDC (weight ≥ 17 kg: 45/200 mg granules; weight < 17 kg: 33.75/150 mg granules) once daily for 12 weeks.
Arm/Group | 3 to < 6 Years Old - LDV/SOF 12 Weeks
Number analyzed (Participants) | 17
percentage of participants
  Did not taste the study drug | 41.2
  Tasted drug with score > 60 to 100 | 17.6
  Tasted drug with score 40 to 60 | 11.8
  Tasted drug with score of 0 to < 40 | 29.4

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs): First dose date up to Week 12 or 24 (depending on group) plus 30 days (includes AEs occurring during the PK Lead-in Phase); All-Cause Mortality: Up to Posttreatment Week 24
Description: Safety Analysis Set included all participants who were enrolled into the study and received at least 1 dose of study drug.
Arm/Group | 12 to < 18 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 12 Weeks | 6 to < 12 Years Old - LDV/SOF 24 Weeks | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks | 3 to < 6 Years Old - LDV/SOF 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/89 | 0/1 | 0/2 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/89 | 0/1 | 0/2 | 0/34
Other Adverse Events (participants affected / at risk) | 62/100 | 54/89 | 1/1 | 2/2 | 22/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12 to < 18 Years Old - LDV/SOF 12 Weeks (N=100) | 6 to < 12 Years Old - LDV/SOF 12 Weeks (N=89) | 6 to < 12 Years Old - LDV/SOF 24 Weeks (N=1) | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks (N=2) | 3 to < 6 Years Old - LDV/SOF 12 Weeks (N=34)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12 to < 18 Years Old - LDV/SOF 12 Weeks (N=100) | 6 to < 12 Years Old - LDV/SOF 12 Weeks (N=89) | 6 to < 12 Years Old - LDV/SOF 24 Weeks (N=1) | 6 to < 12 Years Old - LDV/SOF+RBV 24 Weeks (N=2) | 3 to < 6 Years Old - LDV/SOF 12 Weeks (N=34)
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 14 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 13 | 11 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 11 | 9 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 12 | 12 | 0 | 1 | 8
Fatigue (General disorders) | 13 | 13 | 0 | 1 | 2
Pyrexia (General disorders) | 2 | 15 | 0 | 1 | 7
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 7 | 2 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 3 | 0 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 7 | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 5 | 0 | 0 | 1
Headache (Nervous system disorders) | 26 | 16 | 0 | 1 | 3
Product taste abnormal (Product Issues) | 0 | 0 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 5 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 1 | 1 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0 | 6
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 8 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (8):
  • Study Protocol: Original (2014-07-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/Prot_000.pdf
  • Study Protocol: Amendment 1 (2014-10-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/Prot_001.pdf
  • Study Protocol: Amendment 2 (2014-12-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/Prot_002.pdf
  • Study Protocol: Amendment 3 (2015-05-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/Prot_003.pdf
  • Study Protocol: Amendment 4 (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/Prot_004.pdf
  • Study Protocol: Amendment 5 (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/Prot_005.pdf
  • Study Protocol: Amendment 6 (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/Prot_006.pdf
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT02249182/SAP_007.pdf